CLINICAL TRIAL: NCT01652118
Title: Prophylaxis of Bronchopulmonary Dysplasia With Clarithromycin
Brief Title: Clarithromycin Prophylaxis in Preterm Infants Colonisation With Ureaplasma Urealyticum and Mycoplasma Hominis
Acronym: Claprum
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zekai Tahir Burak Women's Health Research and Education Hospital (Other)
Responsible Party: Principal Investigator, Sadik Yurttutan, Fellowship of neonatology, Zekai Tahir Burak Women's Health Research and Education Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 05059079727
Record Dates: First submitted 2012-07-22; First posted 2012-07-27 (Estimated); Last update posted 2012-07-27 (Estimated); Status verified 2012-07

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: bronchopulmonary dysplasia; clarithromycin; preterm babies
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clarithromycin (Active Comparator): Fist group treated with clarithromycin which is include 10 days application.
  Interventions: Drug: clarithromycin treatment for prophylaxis of bronchopulmonary dysplasia
- placebo (Placebo Comparator): Second group treated with salin as same as amount of clarithromycine volume
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: clarithromycin treatment for prophylaxis of bronchopulmonary dysplasia
  Other Names: Claprum
  Arms: Clarithromycin
Drug: Saline
  Arms: placebo

SUMMARY:
The purpose of this study is to determine of clarithromycin effect on developing of bronchopulmonary dysplasia in preterm babies.

DETAILED DESCRIPTION:
The investigators planned that clarithromycin treatment in preterm babies who are under 1250 grams birth weight.

The investigators aimed with this treatment, the bronchopulmonary dysplasia rate of preterm babies may decrease.

ELIGIBILITY:
Inclusion Criteria:

* all infant must be under 1250 gram birth weight

Exclusion Criteria:

* Major congenital anomaly,
* CardiaC abnormality,
* without inform consent

Ages: 1 Hour to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Bronchopulmonary dysplasia | 28. day of birth
  On the 28. day of birth, The investigator will determine the baby whether has developed bronchopulmonary dysplasia

SECONDARY OUTCOMES:
Overall survival | Participants will be followed for the duration of hospital stay, an expected average of postnatal 40 weeks
  During to hospitalisation the investigator will determine and record some co-morbidities of BPD such as intracranial hemorrhage, necrotizing enterocolitis, patent ductus arteriosus rates.From date of randomization until the end of the hospitalisation up to the 3 months of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ugur Dilmen, Prof. Dr., Study Director — Zekai Tahir Burak Women's Health Research and Education Hospital
Locations (1):
- Zekai Tahir Burak Maternity Teaching Hospital, Ankara, Middle Anatolia, Turkey (Türkiye)